CLINICAL TRIAL: NCT04900675
Title: Effects of Bright Morning Light Exposure on Students' Stress, Mood, Anxiety, Sleep and, Circadian Rest-activity Cycle
Brief Title: Bright Light Intervention to Reduce Students' Stress
Acronym: BLISS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaet Innsbruck (Other)
Collaborators: Bartenbach GmbH (Unknown)
Responsible Party: Principal Investigator, Markus Canazei, Principal Investigator, Universitaet Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 878649
Record Dates: First submitted 2021-04-29; First posted 2021-05-25 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-12

CONDITIONS: Psychological Stress; Physiological Stress; Sleep Disorders, Circadian Rhythm
Keywords: stress; light therapy
MeSH Terms: conditions — Stress, Psychological; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Intervention Model Description: placebo-controlled, randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: After randomisation to the two light intervention study arms, it is only explained to the test persons that the influence of regular exposure to light in the morning is being investigated.
  The control light condition comprises dim, reddish light. The reddish color tone in this light intervention should mask allocation to the study arm. A no-light intervention group (study arm 3) will be established as an additional control condition.
  Data analysis will be carried out by a member of the project team who is blinded to study arm allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- bright white light intervention (Experimental): exposure to 5,000 lux with polychromatic white light with 5,300 Kelvin at eye level; light exposure starts immediately after awakening; light exposure takes place on weekdays (Monday till Friday) over a period of 3 weeks
  Interventions: Other: Bright light intervention
- dim reddish light intervention (Placebo Comparator): exposure to 50 lux with polychromatic reddish light with 2,200 Kelvin at eye level; light exposure starts immediately after awakening; light exposure takes place on weekdays (Monday till Friday) over a period of 3 weeks
  Interventions: Other: Reddish placebo light
- no light intervention (No Intervention): no light intervention takes place in the morning; the study participants follow their natural rhythm of life

INTERVENTIONS:
Other: Bright light intervention — Exposure with 5,000 lux at eye level for one hour and a Correlated Color Temperature of 5,300 Kelvin every morning for three weeks.
  Arms: bright white light intervention
Other: Reddish placebo light — Exposure with 50 lux at eye level for one hour and a Correlated Color Temperature of 2,200 Kelvin every morning for three weeks.
  Arms: dim reddish light intervention

SUMMARY:
Increased stress levels are a significant problem for many students and represent a risk factor for impaired mental and physical health as well as academic performance. Stress levels are particularly high during the preparation phase for major exams.

There is good evidence that light therapy is an effective treatment option to improve mood in affective disorders.

The present study aims at investigating the psychophysiological effects of a 3-week morning bright light exposure in reducing stress and stress-related problems in students preparing for major exams.

DETAILED DESCRIPTION:
Increased students' stress represents a significant risk factor for impaired mental and physical health as well as academic performance. The World Mental Health Survey (WHO) reports a 12-month prevalence of mental illness of 20.3% among students, with anxiety disorders (14.7%), affective disorders (9.9%), and substance abuse (6.7%) being particularly prominent. Moreover, six out of 10 students suffer from impaired sleep quality.

Offering an effective treatment for stress-related symptoms in students is a challenge. In situations of intense stress, conventional methods such as relaxation and mindfulness-based programs often fail because of poor prior practice. Only a few students apply cognitive behavioral interventions. Although medication might decrease stress symptoms within days, the side effects of drugs cannot be ignored. Therefore, there is a need for effective and efficient treatment of acute stress symptoms in students.

Bright light therapy is an effective treatment for several mental disorders, e.g. affective disorders and sleep disorders. There is some evidence, that exposure to bright light may even reduce stress in patients with burnout symptoms. Thus, exposure to bright light may be a promising new option to reduce academic stress and improve mood and sleep parameters.

In the present study, a large-area desk lamp, which emits diffuse light and is controllable in its luminance and correlated color temperature is used. Study participants are randomly assigned to one of three study arms: (i) exposure to polychromatic light of 5,000 lux and 5,300 Kelvin, (ii) exposure to polychromatic light of 50 lux and 2,200 Kelvin, or (iii) no light intervention. Data collection takes place in winter periods.

ELIGIBILITY:
Inclusion Criteria:

* students from the faculty of medicine, pharmacy, and law
* major exam at least 5 weeks ahead
* major depressive disorder (PHQ-9): Score > 4
* possession of smartphone and data plan

Exclusion Criteria:

* suicidal ideation (BDI, Item i): Rating > 1
* seasonal affective disorder (PIDS-A): Score > 11
* taking medication which increases photo-sensitivity
* taking medication to increase cognitive performance
* starting or changing pharmacotherapy for affective disorders and anxiety disorders within the last two weeks
* changing of all kinds of medication within the last two weeks
* headache (PHQ-D, Item f): Rating "severly impaired"
* increased light sensitivity: Item "Wearing sunglasses outside on sunny days" is answered with 'often' or 'very often'
* currently undergoing psychotherapeutic treatment
* the presence of an eye disease for which light therapy is contraindicated

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
subjective stress level - baseline/post | Change from baseline PSS-10 sum score at the end of week 3
  Perceived Stress Scale (PSS-10); scale: PSS-10 sum score; range:0 - 40; higher scores mean a higher subjective stress level
subjective stress level - baseline/post | Change from baseline PSQ-20 sum score at the end of week 3
  Perceived Stress Questionnaire (PSQ-20); scale: PSQ-20 sum score; range: 20 - 80; higher scores mean a higher subjective stress level
subjective stress level - on weekdays | Change of daily PSQ-20 sum score at each weekday during the light intervention period up to 3 weeks
  Perceived Stress Questionnaire (PSQ-20); scale: PSQ-20 sum score; range: 20 - 80; higher scores mean a higher subjective stress level

SECONDARY OUTCOMES:
anxiety | Change from baseline STAI-trait sum score at the end of week 3
  State-Trait Anxiety Inventory (STAI - form Y) - 20 trait items; scale: STAI-trait sum score; range: 20 - 80; higher scores mean a higher subjective anxiety level
mood | Change from baseline CES-D sum score at the end of week 3
  Center for Epidemiologic Studies Depression Scale (CES--D); scale: CES-D sum score; range: 0 - 60; higher scores mean a higher subjective depression level
sleep quality | Change from baseline global PSQI score at the end of week 3
  Pittsburgh Sleep Quality Index (PSQI); scale: global PSQI score; range: 0 - 21; higher scores mean a lower subjective sleep quality
sleep quality - total sleep time | Change of TST at each night during the light intervention period up to 3 weeks
  Wrist actimetry to measure daily total sleep time (TST); scale: sleep duration; range: >0 (minutes); higher TST means longer sleep period
sleep quality - sleep onset latency | change of SOL at each night during the light intervention period up to 3 weeks
  Wrist actimetry to measure daily sleep onset latency (SOL); scale: duration to fall asleep; range: >0 (minutes); higher SOL means longer period to fall asleep
sleep quality - wake after sleep onset | change of WASO at each night during the light intervention period up to 3 weeks
  Wrist actimetry to measure daily wake after sleep onset (WASO); scale: duration of being awake during sleep period; range: greater than or equal to 0 (minutes); higher WASO means longer wake periods after sleep onset
sleep quality - sleep efficiency | change of SE at each night during the light intervention period up to 3 weeks
  Wrist actimetry to measure daily sleep efficiency (SE); scale: percentage; range: 0 - 100; higher SE means a higher undisturbed sleep
circadian rest/activity rhythm - interdaily stability | change of IV at each of the three light intervention weeks up to 3 weeks
  Circadian rest-activity cycle parameter interdaily stability (IS) derived from weekly wrist actimetry data; scale: real number; range: 0 -1; higher IS means a higher stability in daily rest-activity cycles
circadian rest/activity rhythm - intradaily variability | change of IS at each of the three light intervention weeks up to 3 weeks
  Circadian rest-activity cycle parameter intradaily variability (IV) derived from averaged wrist actimetry data over a period of 1 week; scale: real number; range: 0 - 2; higher IV means a higher variability in 24-h rest-activity cycle
physiological stress reaction | Change from baseline hair cortisol level at the end of week 3
  cortisol level measured from hair sample; scale: real number (pg/mg); range: >0; higher hair cortisol level means higher physiological stress
adverse effects - short-term | day 5
  astenopic complaints measured with 12 items; scale: sum score; range: 10 - 60; higher sum score means more astenopic complaints
adverse effects - long-term | day 15
  astenopic complaints scale measured with 12 items: sum score; range: 10 - 60; higher sum score means more astenopic complaints

OTHER OUTCOMES:
resilience | Change from baseline RS-11 sum score at the end of week 3
  Resilience Scale (RS-11); scale: RS-11 sum score; range: 11 - 77; higher RS-11 sum score means more perceived resilience
stress coping | Change from baseline multidimensional CISS scale at the end of week 3
  Coping Inventory for Stressful Situations (CISS) - 24 items; three-dimensional CISS scale: (a) task-oriented coping; (b) emotion-oriented coping, and (c) avoidance-oriented coping; range for each dimension: 8 - 40; higher score in each dimension means higher preference for particular stress coping style
learning strategies | Change from baseline multidimensional LIST-K scale at the end of week 3
  Learning Strategies of University Students (LIST-K) - 36 items; multidimensional LIST-K scale: 13 subscales; range for each dimension: 3 - 15; higher score in each dimension means higher preference for particular learning strategy
psychological distress | Change from baseline BSI-18 overall score at the end of week 3
  Brief Symptom Inventory (BSI-18); scale: BSI-18 sum score; range: 18 - 90; higher BSI-18 sum score means higher psychological distress
somatic symptoms | Change from baseline SSS-8 sum score at the end of week 3
  The somatic symptom scale (SSS-8); scale: SSS-8 sum score; range: 0 - 32; higher SSS-8 sum score means higher somatic complaints
satisfaction with light intervention - short-term | day 5
  2 items: (a) recommendation of light intervention to a friend and (b) follow-up usage of light intervention for own purposes; scale: binary score ('yes', 'no'); range: 0 - 1; higher binary scores indicate recommendation and follow-up usage of the light intervention
satisfaction with light intervention - long-term | day 15
  2 items: (a) recommendation of light intervention to a friend and (b) follow-up usage of light intervention for own purposes; scale: binary score ('yes', 'no'); range: 0 - 1; higher binary scores indicate recommendation and follow-up usage of the light intervention
daily mood state | changes from before the light intervention of the two-dimensional PANAS scale at the end of light intervention at each weekday during the light intervention period up to 3 weeks
  Positive and Negative Affect Schedule (PANAS); two-dimensional PANAS scale: sum score for positive and negative mood state; range for each dimension: 10 - 50; higher PANAS scores mean higher positive and negative mood state, respectively
weekly social rhythms | changes in SRM scores in week 1, week 2, and week 3
  The Social Rhythm Metric (SRM) measures the regularity in the occurance of 17 daily events; scale: SRM score; range: 0 - 7; higher SRM scores mean more regular occurance of daily events
anxiety state | changes from before the light intervention STAI-state sum score at the end of light intervention in week 1, week 2, and week 3
  State-Trait Anxiety Inventory (STAI - form Y) - 20 state items; scale: STAI-state sum score; range: 20 - 80; higher scores mean a higher subjective current anxiety level
cognitive performance | changes from before the light intervention NLT number of correct answers at the end of light intervention in week 1, week 2, and week 3
  The Number Letter Task (NLT) measures task switching performance; scale: number of correct answers; range: integer greater than or equal to 0; higher NLT scores means a better task switching performance
exam anxiety | changes of multidimensional PAF scale at week 1, week 2, and week 3
  German Test Anxiety Inventory (PAF); four-dimensional PAF scale: (a) excitement, (b) concern, (c) interference, and (d) lack of confidence; range for each dimension: 5 - 20; higher scale means higher test anxiety in the corresponding dimension

CONTACTS AND LOCATIONS:
Overall Officials: Markus Canazei, PhD, Principal Investigator — University of Innsbruck
Locations (1):
- University of Innsbruck, Innsbruck, Tyrol, Austria